CLINICAL TRIAL: NCT06275867
Title: The Impact of Access to Higher-quality Care Services on Health-seeking Patterns
Brief Title: Improved Access to Quality Care and Healthcare Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SOPRIMA//T023635
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-02

CONDITIONS: Health Care Utilization; Health Knowledge, Attitudes, Practice; Health, Subjective
MeSH Terms: conditions — Patient Acceptance of Health Care; Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): In this group, participants will have free access to government facilities (usual care)
- Convenient group (Experimental): In this group, for the duration of the study, participants will be given free access to a small number of private providers located relatively close by (less than 30 minutes).
  Interventions: Other: Free high-quality care; Other: Close distance
- Inconvenient group (Experimental): In this group, for the duration of the study, participants will be given free access to a small number of private providers located relatively far (about one hour).
  Interventions: Other: Free high-quality care; Other: Far distance

INTERVENTIONS:
Other: Free high-quality care — Participants are able to take their child to receive free consultations and treatment in a network of contracted private healthcare providers.
  Arms: Convenient group; Inconvenient group
Other: Close distance — The network of contracted providers is located close to where participants live.
  Arms: Convenient group
Other: Far distance — The network of contracted providers is located far to where participants live.
  Arms: Inconvenient group

SUMMARY:
This study is an individual-level randomised controlled trial which looks at the effect of providing free access to higher quality providers in urban South Africa. The study will recruit about 1,500 individuals with a child aged 5 or under. They will be randomly allocate to a control group (CONTROL) with the default free access to government facilities or one of the two treatment groups where they will have free access to private providers located either relatively close (CONVENIENT) by or relatively far (INCONVENIENT). The primary outcomes be overuse and underuse of healthcare services for children under 5

DETAILED DESCRIPTION:
In many low-income settings, provision of social services by the public sector is plagued by problems of quality and low accountability to users. As a result, low expected benefits or fear of neglect by service providers may delay the use of needed services, even when those are free.

In South Africa, the health system is characterised by stark inequalities, with most of the population only able to seek care in free government facilities. The low quality of the public sector, where patients wait long times to be seen by nurses, is believed to lead many to delay needed care and prevent health outcome improvement. The government of South Africa is developing proposals to introduce a national health insurance scheme that would provide free access to private providers who deliver higher care quality. However, concerns about the unequal geographical distribution of private providers raise questions about the potential benefits of the reform. This study asks several questions to inform this reform:

1. Does access to higher-quality care reduce under-use of services for children but also increase overuse?
2. Does access to higher-quality care lead to improved health knowledge of parents and better health outcomes for children?
3. Are these effects mitigated by the distance to the contracted providers? A randomised controlled trial is used to answer these questions. The study will recruit about 1,500 individuals who are the primary caregiver of at least one child aged six or under. and randomly allocate them to a control group (CONTROL) with the default free access to government facilities or one of the two treatment groups where they will have free access to private providers located either relatively close (CONVENIENT) by or relatively far (INCONVENIENT).

The primary outcomes will be the proportion of visits that are considered unnecessary (overuse) and the number of days of illness where care-seeking is recommended by guidelines but not sought by the child's parent or guardian.

Secondary outcomes will include (1) the number of days with ill-health symptoms; (2) out-of-pocket expenditures; (3) health knowledge of parents; (4) subjective and (5) objective measures of child's health.

ELIGIBILITY:
Inclusion Criteria:

* parent has a child aged under 6 years old and over 2 months old

Exclusion Criteria:

* is planning to move out of the area in the next 3 months
* has private medical aid

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Underuse | 12 weeks
  number of days of illness where care-seeking is recommended by guidelines but not sought by the child's parent or guardian
Overuse | 12 weeks
  proportion of primary health care visits that are considered unnecessary

SECONDARY OUTCOMES:
Illness duration | 12 weeks
  number of days with ill-health symptoms
Out-of-pocket expenditures | 12 weeks
  Direct (consultations, drugs) and indirect (transport) expenditures spent on health care
Health knowledge | Endline survey (i.e. 12 weeks approximately after the start of the intervention)
  Index of knowledge of parents in relation to preventive and curative care. Parents will answer as series of knowledge questions relative to care-seeking patterns for children (with correct and incorrect responses). For each individual, a score will be computing by adding up all of the correct responses (1 point per correct response, 0 for incorrect), so a higher score will reflect a better knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Mylene Lagarde, PhD, Principal Investigator — London School of Economics and Political Science
Locations (1):
- HDSS Soweto clusters, Soweto, Gauteng, South Africa